CLINICAL TRIAL: NCT05250115
Title: This is a Prospective, Single-arm, Multicenter, Observational Non-interventional Study (NIS) in Germany of Patient Characteristics, Usage, and Effectiveness of Abrocitinib in Patients With Moderate to Severe Atopic Dermatitis (AD)
Brief Title: A Study to Learn About Abrocitinib in Adult Patients With Moderate to Severe Atopic Dermatitis
Status: Terminated | Type: Observational
Why Stopped: Business decision: Due to the slow recruitment, the sponsor decided to discontinue the study early.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7451089; ABROAD (Other: Alias Study Number)
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic Dermatitis; Abrocitinib; JAK inhibitors
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Evaluate the effectiveness, usage and patient characteristics of real-world use of Abrocitinib: This is a 60-month, prospective, non-interventional, multicenter study to evaluate the effectiveness, usage and patient characteristics of abrocitinib in patients with moderate to severe AD in a real-world setting.
  Eligible patients will be followed up from the date of first Abrocitinib prescription for 12 months. from the date of enrollment. Patients who are switched from the initial abrocitinib therapy to other therapies continue to be observed. Patient documentation is expected quarterly as per standard clinical practice.

SUMMARY:
The purpose of this non-interventional observational study is to learn about the safety and effects of the medicinal product (called Abrocitinib) for the potential treatment of moderate to severe atopic dermatitis (AD). AD is a long-lasting disease that causes redness and irritation of the skin. This non-interventional study is seeking participants who is eligible for Abrocitinib treatment according to the summary of product characteristics (SmPC):

* Are aged at least 18 years old
* Have a confirmed diagnosis of AD by a skin doctor
* Decide to start treatment with Abrocitinib as part of routine clinical practice
* Have a personally signed and dated informed consent document. This is used to indicate that the patient has been informed of all pertinent aspects of the study and data privacy aspects

Participants will take the medicinal product as prescribed in the real-world setting. We will examine the experiences of people receiving Abrocitinib. This will help us determine if the medicinal product is effective and safe. Participants will take part in this study for 3 months. During this time, participants will be followed up from the date of their first Abrocitinib prescription for 12 months. During this non-interventional study, some participants may switch to other therapies after their initial Abrocitinib therapy. We will follow these participants further when they switch therapy to monitor their experiences. Participant documentation is expected quarterly as per standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Confirmed diagnosis of AD by dermatologist prior to study inclusion
* Patient for whom the decision to initiate treatment with abrocitinib was made as part of routine clinical practice irrespective of the patients being

  1. abrocitinib naive or,
  2. patients who reinitialize treatment with abrocitinib after being off treatment for ≥28 days prior to study inclusion
* Patient is eligible for abrocitinib treatment according to Summary of Product Characteristics (SmPC)
* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the non-interventional study

Exclusion Criteria:

* Contraindications according to SmPC
* Receipt of any investigational drug within 3 months or longer if required according to wash-out period prior to inclusion or participation in a clinical trial during observation period
* Patients being treated with abrocitinib within a time period of <28 days prior to the timepoint of study inclusion
* Patients who are investigational site staff members or patients who are Pfizer employees directly involved in the conduct of the non-interventional study
* Patients who are unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A prospective, single-arm, multi-center, observational non-interventional study looking at adult patients with moderate-severe atopic dermatitis, who have been chosen to start treatment with Abrocitinib in Germany according to the current routine practice of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- Germany (38):
  - Elbe Kliniken Stade - Buxtehude GmbH, Buxtehude, Lower Saxony
  - ÜUeberoertliche Gemeinschaftspraxis Jost Kai Rietkoetter Robert Jablonka, Gelsenkirchen, North Rhine-Westphalia
  - Dermatologische Gemeinschaftspraxis Dres. Quist PartG, Mainz, Rhineland-Palatinate
  - "Magdeburger company for Medical studies & Services", Magdeburg, Saxony-Anhalt
  - Hautärztliche Gemeinschaftspraxis, Ahaus
  - Hautarztpraxis Dr. Virgil Mihaescu, Augsburg
  - Dermatologie Bad Kreuznach - Dr. med. Georg Mauer, Bad Kreuznach
  - Praxis Dr. A. Magerl, Bensheim
  - Hautzentrum, Bergen
  - Dr. Christiane Handrick Hautarztpraxis, Berlin
  - Dres. Ziethen-Stavermann GbR, Berlin
  - Hautarztpraxis Dr. med. Thomas Schirmer, Berlin
  - Hautzentrum Weißensee, Berlin
  - Hautarztpraxis Weid, Bingen
  - Hautarztpraxis an der Hase Studienzentrum, Bramsche
  - Hautärzte Braunschweig, Braunschweig
  - Hautarztpraxis Dr. med. Daniela Kasche, Buxtehude
  - Praxis Dr. Voth, Cologne
  - BAG Freitag und Knöll, Falkensee
  - Haut- und Laserzentrum Freisung Prof. Kurzen, Freising
  - Hautarztpraxis Dr. med Michael Loth, Gernsbach
  - Hautarztpraxis Dr. Brinkmann, Schult & Samimi-Fard, Gladbeck
  - Cutaneum Praxis Dr. Buck, Hamburg
  - Hautarztpraxis Dr. med. Matthias Lütten, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - dermaSANA, Karlsruhe
  - Kosmedikulm, Kulmbach
  - Dr. Beate Schwarz, Langenau
  - Dermatologie Mölln, Praxis Dr Segert, Mölln
  - ZENTderma, Dr. Rolf Ostendorf, Mönchengladbach
  - Hautarztpraxis Dorittke / Kardorff, Mönchengladbach
  - Hautarztpraxis Dr. Susanne Gißler-Walter, Mutterstadt
  - Praxis Dr. Quack, München
  - Dermatologische Praxis im Hautzentrum Johannis Dr. med. Esther Völkel, Nuremberg
  - Hautarztpraxis Mortazawi, Remscheid
  - Dermatologische Spezialpraxis Dr. med. Ralph von Kiedrowski, Selters
  - Dermatologisches Studienzentrum Hunsrück - DSH, Simmern
  - Hautarztpraxis Dr. Hoffmann, Witten

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451089

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 112 participants who were diagnosed with moderate to severe atopic dermatitis (AD) and received abrocitinib treatment were included, of which 2 participants violated the inclusion/exclusion criteria, and a total 110 participants were included in the full analysis set (FAS). Participants were followed up for 12 months.
Groups:
- Abrocitinib: Participants with moderate to severe AD who received treatment with oral abrocitinib in a real-world setting were observed in this prospective study.
Period: Overall Study
Arm/Group | Abrocitinib
Started | 110
Completed | 41
Not Completed | 69
Not completed — Premature study end | 40
Not completed — Adverse Event | 8
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 6
Not completed — Withdrawal of informed consent | 1
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all participants with informed consent who met the eligibility criteria and received at least one dose of abrocitinib.
Groups:
- Abrocitinib: Participants with moderate to severe AD who received treatment with oral abrocitinib were observed in this prospective study.
Arm/Group | Abrocitinib
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.59 (15.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: All participants who consented to disclose their ethnicity details.
  Participants
    Ethnicity: number analyzed (Participants) | 95
    Ethnicity: Caucasian | 86
    Ethnicity: Non-Caucasian | 2
    Ethnicity: Unknown | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Investigator's Global Assessment (IGA) Score of Clear (0) or Almost Clear (1) at Month 3
Description: The IGA is a tool used to assess the severity of AD (excluding scalp, palms and soles) on a 5-point scale that ranges from 0 to 4, where 0 indicates clear (no signs of AD), 1 indicates almost clear (minimal signs of AD), 2 indicates mild AD, 3 indicates moderate AD and 4 indicates severe AD, higher scores indicated greater severity of AD. Percentage of participants with score of "Clear" (score 0) or "Almost Clear" (score 1) according to IGA were reported in this outcome measure.
Time Frame: At Month 3
Population: The FAS included all participants with informed consent who met the eligibility criteria and received at least one dose of abrocitinib. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Abrocitinib
Number analyzed (Participants) | 84
Percentage of participants | 35.71

2. Primary Outcome: Percentage of Participants With 75% Reduction From Baseline in Eczema Area and Severity Index (EASI) at Month 3
Description: The EASI assessed both clinical signs of AD as well as extent of disease. For body regions such as "head and neck", "trunk", "upper extremities" and "lower extremities" the extent of eczema was assessed by an area score between 0 (0% of body surface area [BSA] affected) and 6 (90 to 100% of BSA affected), respectively. For each area the severity of clinical signs of AD such as "erythema", "edema/papulation", "excoriation" and "lichenification" were scored from 0 to 3, respectively where 0= absent; 1= mild; 2= moderate; 3= severe. The scores for the signs were added for each area and multiplied by the respective area score. The EASI for an individual was calculated as weighted sum: 0.1*score for head/neck + 0.3*score for trunk + 0.2*score for upper extremities + 0.4*score for lower extremities. The total score ranged from 0 to 72, higher scores represented greater severity of AD. EASI 75 response was defined as at least a 75% reduction in EASI relative to baseline.
Time Frame: At Month 3
Population: FAS included all participants with informed consent who met the eligibility criteria and received at least one dose of abrocitinib. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Abrocitinib
Number analyzed (Participants) | 84
Percentage of participants | 47.62

3. Secondary Outcome: Percentage of Participants Who Achieved IGA Score of Clear (0) or Almost Clear (1) Until End of Study
Description: The IGA is a tool used to assess the severity of AD (excluding scalp, palms and soles) on a 5-point scale that typically ranges from 0 to 4, where 0 indicates clear (no signs of AD), 1 indicates almost clear (minimal signs of AD), 2 indicates mild AD, 3 indicates moderate AD and 4 indicates severe AD, higher scores indicated greater severity of AD. Percentage of participants with score of "Clear" (score 0) or "Almost Clear" (score 1) according to IGA were reported in this outcome measure.
Time Frame: From Baseline (Day 1) up to end of study (Month 12)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Abrocitinib
Number analyzed (Participants) | 101
Percentage of participants | 51.49

4. Secondary Outcome: Percentage of Participants With 75% Reduction From Baseline in EASI Score Until End of Study
Description: The EASI assessed both clinical signs of AD as well as extent of disease. For body regions such as "head and neck", "trunk", "upper extremities" and "lower extremities" the extent of eczema was assessed by an area score between 0 (0% of BSA affected) and 6 (90 to 100% of BSA affected), respectively. For each area the severity of clinical signs of AD such as "erythema", "edema/papulation", "excoriation" and "lichenification" were scored from 0 to 3, respectively where 0= absent; 1= mild; 2= moderate; 3= severe. The scores for the signs were added for each area and multiplied by the respective area score. The EASI for an individual was calculated as weighted sum: 0.1*score for head/neck + 0.3*score for trunk + 0.2*score for upper extremities + 0.4*score for lower extremities. The total score ranged from 0 to 72, higher scores represented greater severity of AD. EASI 75 response was defined as at least a 75% reduction in EASI relative to baseline.
Time Frame: From Baseline (Day 1) up to end of study (Month 12)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Abrocitinib
Number analyzed (Participants) | 101
Percentage of participants | 63.37

5. Secondary Outcome: Percentage of Participants With 90% Reduction From Baseline in EASI Score Until End of Study
Description: The EASI assessed both clinical signs of AD as well as extent of disease. For body regions such as "head and neck", "trunk", "upper extremities" and "lower extremities" the extent of eczema was assessed by an area score between 0 (0% of BSA affected) and 6 (90 to 100% of BSA affected), respectively. For each area the severity of clinical signs of AD such as "erythema", "edema/papulation", "excoriation" and "lichenification" were scored from 0 to 3, respectively where 0= absent; 1= mild; 2= moderate; 3= severe. The scores for the signs were added for each area and multiplied by the respective area score. The EASI for an individual was calculated as weighted sum: 0.1*score for head/neck + 0.3*score for trunk + 0.2*score for upper extremities + 0.4*score for lower extremities. The total score ranged from 0 to 72, higher scores represented greater severity of AD. EASI 90 response was defined as at least a 90% reduction in EASI relative to baseline.
Time Frame: From Baseline (Day 1) up to end of study (Month 12)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Abrocitinib
Number analyzed (Participants) | 101
Percentage of participants | 42.57

6. Secondary Outcome: Percentage of Participants Who Achieved IGA Score of Clear (0) or Almost Clear (1) and a Reduction of >= 2 Points From Baseline Until End of Study
Description: The IGA is a tool used to assess the severity of AD (excluding scalp, palms and soles) on a 5-point scale that typically ranges from 0 to 4, where 0 indicates clear (no signs of AD), 1 indicates almost clear (minimal signs of AD), 2 indicates mild AD, 3 indicates moderate AD and 4 indicates severe AD, higher scores indicated greater severity of AD. Percentage of participants with score of "Clear" (score 0) or "Almost Clear" (score 1) and a reduction of >=2 points from baseline according to IGA were reported in this outcome measure.
Time Frame: From Baseline (Day 1) up to end of study (Month 12)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Abrocitinib
Number analyzed (Participants) | 101
Percentage of participants | 47.52

7. Secondary Outcome: Percentage Change From Baseline in IGA Total Score at Months 1, 3, 6, 9 and 12
Description: The IGA is a tool used to assess the severity of AD (excluding scalp, palms and soles) on a 5-point scale that typically ranges from 0 to 4, where 0 indicates clear (no signs of AD), 1 indicates almost clear (minimal signs of AD), 2 indicates mild AD, 3 indicates moderate AD and 4 indicates severe AD, higher scores indicated greater severity of AD.
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: FAS included all participants with informed consent who met the eligibility criteria and received at least one dose of abrocitinib. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Abrocitinib
Number analyzed (Participants) | 81
Percentage change
  Month 1 | -38.79 (33.55)
  Month 3: number analyzed (Participants) | 67
  Month 3 | -50.37 (31.06)
  Month 6: number analyzed (Participants) | 57
  Month 6 | -46.05 (33.15)
  Month 9: number analyzed (Participants) | 44
  Month 9 | -41.86 (32.07)
  Month 12: number analyzed (Participants) | 34
  Month 12 | -38.97 (40.45)

8. Secondary Outcome: Percentage Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Total Score at Months 1, 3, 6, 9 and 12
Description: SCORAD total score was a validated scoring index for AD that assessed severity by combining A: extent, B: severity and C: subjective symptoms. A: a rule of 9 was used to calculate BSA affected by AD as a % of whole-BSA for each body region- head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; 1% for genitals. Score for each body region was added to determine A (0-100). B: severity of each sign (erythema; edema; oozing; excoriation; lichenification; dryness) was assessed as none =0, mild =1, moderate =2, severe =3, severity scores were added to give B (0-18). C: based on itching and sleep deprivation, each scored (0-10) where, 0= no itch/no sleeplessness and 10= worst imaginable itch/sleeplessness, scores for itch and sleeplessness were added to give C (0-20). The total score for an individual was calculated as A/5 + 7B/2 + C and ranged from 0-103; higher SCORAD scores = greater severity of AD.
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Abrocitinib
Number analyzed (Participants) | 71
Percentage change
  Month 1 | -48.53 (28.43)
  Month 3: number analyzed (Participants) | 59
  Month 3 | -50.60 (27.60)
  Month 6: number analyzed (Participants) | 44
  Month 6 | -53.41 (29.64)
  Month 9: number analyzed (Participants) | 34
  Month 9 | -43.46 (31.86)
  Month 12: number analyzed (Participants) | 28
  Month 12 | -50.08 (30.81)

9. Secondary Outcome: Absolute EASI Total Score at Months 1, 3, 6, 9 and 12
Description: The EASI assessed both clinical signs of AD as well as extent of disease. For body regions such as "head and neck", "trunk", "upper extremities" and "lower extremities" the extent of eczema was assessed by an area score between 0 (0% of BSA affected) and 6 (90 to 100% of BSA affected), respectively. For each area the severity of clinical signs of AD such as "erythema", "edema/papulation", "excoriation" and "lichenification" were scored from 0 to 3, respectively where 0= absent; 1= mild; 2= moderate; 3= severe. The scores for the signs were added for each area and multiplied by the respective area score. The EASI for an individual was calculated as weighted sum: 0.1*score for head/neck + 0.3*score for trunk + 0.2*score for upper extremities + 0.4*score for lower extremities. The total score ranged from 0 to 72, higher scores represented greater severity of AD.
Time Frame: At Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abrocitinib
Number analyzed (Participants) | 85
Units on a scale
  Month 1 | 5.09 (6.57)
  Month 3: number analyzed (Participants) | 69
  Month 3 | 4.37 (7.03)
  Month 6: number analyzed (Participants) | 56
  Month 6 | 3.65 (4.50)
  Month 9: number analyzed (Participants) | 45
  Month 9 | 4.70 (5.47)
  Month 12: number analyzed (Participants) | 33
  Month 12 | 5.11 (8.09)

10. Secondary Outcome: Percentage Change From Baseline in EASI Total Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 9
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Abrocitinib
Number analyzed (Participants) | 84
Percentage change
  Month 1 | -57.00 (64.37)
  Month 3: number analyzed (Participants) | 69
  Month 3 | -70.11 (31.71)
  Month 6: number analyzed (Participants) | 55
  Month 6 | -67.89 (47.82)
  Month 9: number analyzed (Participants) | 45
  Month 9 | -69.16 (32.03)
  Month 12: number analyzed (Participants) | 33
  Month 12 | -71.58 (35.79)

11. Secondary Outcome: Absolute Change From Baseline in IGA Total Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 7
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abrocitinib
Number analyzed (Participants) | 81
Units on a scale
  Month 1 | -1.31 (1.16)
  Month 3: number analyzed (Participants) | 67
  Month 3 | -1.66 (1.11)
  Month 6: number analyzed (Participants) | 57
  Month 6 | -1.51 (1.12)
  Month 9: number analyzed (Participants) | 44
  Month 9 | -1.39 (1.06)
  Month 12: number analyzed (Participants) | 34
  Month 12 | -1.38 (1.30)

12. Secondary Outcome: Percentage of Participants Who Achieved at Least 4 Point Improvement on Pruritus Numerical Rating Scale (NRS) From Baseline Until End of Study
Description: The pruritus-NRS comprised of one item and the score ranged from 0 ("no itch") to 10 ("worst imaginable itch"). Higher scores indicated greater severity. Participants were asked to rate the intensity of their average pruritus using this scale. Percentage of participants who achieved at least 4-point improvement on pruritus NRS are reported in this outcome measure.
Time Frame: From Baseline (Day 1) up to end of study (Month 12)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Abrocitinib
Number analyzed (Participants) | 101
Percentage of participants | 42.57

13. Secondary Outcome: Percentage of Participants With Pruritus NRS Score Less Than or Equal to (<=1)
Description: The pruritus-NRS was comprised of one item and the score ranged from 0 ("no itch") to 10 ("worst imaginable itch"). Higher scores indicated greater severity. Participants were asked to rate the intensity of their average pruritus using this scale. Percentage of participants with pruritus NRS score <=1 are reported in this outcome measure.
Time Frame: From Baseline (Day 1) up to end of study (Month 12)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Abrocitinib
Number analyzed (Participants) | 101
Percentage of participants | 29.70

14. Secondary Outcome: Percentage Change From Baseline in Peak-Pruritus (PP) NRS at Months 1, 3, 6, 9 and 12
Description: PP NRS evaluated itching in the last 24 hours on a scale ranging from no itching (0) to worst possible itching (10). Higher scores indicated greater severity.
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Abrocitinib
Number analyzed (Participants) | 59
Percentage change
  Month 1 | -53.15 (36.81)
  Month 3: number analyzed (Participants) | 36
  Month 3 | -43.17 (39.01)
  Month 6: number analyzed (Participants) | 40
  Month 6 | -48.41 (47.88)
  Month 9: number analyzed (Participants) | 34
  Month 9 | -39.11 (74.06)
  Month 12: number analyzed (Participants) | 27
  Month 12 | -37.41 (65.89)

15. Secondary Outcome: Percentage Change From Baseline in Patient Oriented Eczema Measure (POEM) Score at Months 1, 3, 6, 9 and 12
Description: POEM was a participant-reported measure that assessed AD symptoms. The participants self-evaluated the frequency of occurrence and severity of 7 symptoms (such as itching and burning of the skin) within the last week, each according to a 5-point Likert scale from 0 ("at no day") to 4 ("at all days"). The total POEM score was summed over the symptoms and ranged from 0 (clear) to 28 points (very severe), where higher score indicated greater severity.
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Abrocitinib
Number analyzed (Participants) | 58
Percentage change
  Month 1 | -54.53 (35.86)
  Month 3: number analyzed (Participants) | 34
  Month 3 | -49.90 (39.39)
  Month 6: number analyzed (Participants) | 38
  Month 6 | -49.54 (38.25)
  Month 9: number analyzed (Participants) | 34
  Month 9 | -42.42 (45.50)
  Month 12: number analyzed (Participants) | 23
  Month 12 | -44.74 (63.31)

16. Secondary Outcome: Percentage Change From Baseline in Medical Outcomes Study Sleep (MOS) Scale at Months 1, 3, 6, 9 and 12
Description: The MOS-Sleep Scale is a self-administered questionnaire consisting of 12 items that assess key constructs of sleep. Instrument scoring yields 7 subscales (sleep disturbance, snoring, Sleep short of breath and headache, sleep quantity (raw scores), optimal sleep, sleep adequacy, and sleep somnolence) as well as sleep problems index I and II and all have score ranges from 0 (no sleep problems) to 100 (greater sleep problems), where higher scores indicated more sleep problems, with exception of sleep adequacy which was scored as 0 (least sleep adequacy) to 100 (better sleep adequacy) where higher scores indicated higher sleep adequacy, and optimal sleep scored as 0 (less quantity of sleep) to 24 (greater quantity of sleep), where higher scores indicated higher quantity sleep.
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Abrocitinib
Number analyzed (Participants) | 65
Percentage change
  Month 1: Sleep disturbance: number analyzed (Participants) | 64
  Month 1: Sleep disturbance | -30.42 (40.76)
  Month 1: Snoring: number analyzed (Participants) | 48
  Month 1: Snoring | -15.80 (52.09)
  Month 1: Sleep short of breath and headache: number analyzed (Participants) | 27
  Month 1: Sleep short of breath and headache | -34.57 (51.46)
  Month 1: Sleep Adequacy: number analyzed (Participants) | 60
  Month 1: Sleep Adequacy | 46.52 (108.77)
  Month 1: Sleep Somnolence: number analyzed (Participants) | 61
  Month 1: Sleep Somnolence | -14.23 (56.05)
  Month 1: Sleep Quantity (raw scores): number analyzed (Participants) | 57
  Month 1: Sleep Quantity (raw scores) | 13.94 (39.40)
  Month 1: Optimal Sleep Scale: number analyzed (Participants) | 18
  Month 1: Optimal Sleep Scale | -27.78 (46.09)
  Month 1: Sleep Problems Index I: number analyzed (Participants) | 64
  Month 1: Sleep Problems Index I | -15.45 (56.08)
  Month 1: Sleep Problems Index II | -20.91 (39.67)
  Month 3: Sleep Disturbance: number analyzed (Participants) | 37
  Month 3: Sleep Disturbance | -39.93 (31.15)
  Month 3: Snoring: number analyzed (Participants) | 30
  Month 3: Snoring | -13.61 (52.77)
  Month 3: Sleep short of breath and headache: number analyzed (Participants) | 17
  Month 3: Sleep short of breath and headache | -54.90 (46.68)
  Month 3: Sleep Adequacy: number analyzed (Participants) | 34
  Month 3: Sleep Adequacy | 81.69 (141.71)
  Month 3: Sleep Somnolence: number analyzed (Participants) | 38
  Month 3: Sleep Somnolence | -15.71 (68.76)
  Month 3: Sleep Quantity (raw scores): number analyzed (Participants) | 31
  Month 3: Sleep Quantity (raw scores) | 23.31 (48.74)
  Month 3: Optimal Sleep Scale: number analyzed (Participants) | 8
  Month 3: Optimal Sleep Scale | -12.50 (35.36)
  Month 3: Sleep Problems Index I: number analyzed (Participants) | 38
  Month 3: Sleep Problems Index I | -33.27 (30.21)
  Month 3: Sleep Problems Index II: number analyzed (Participants) | 38
  Month 3: Sleep Problems Index II | -34.49 (25.42)
  Month 6: Sleep Disturbance: number analyzed (Participants) | 41
  Month 6: Sleep Disturbance | -32.02 (52.68)
  Month 6: Snoring: number analyzed (Participants) | 36
  Month 6: Snoring | -8.10 (63.01)
  Month 6: Sleep short of breath and headache: number analyzed (Participants) | 18
  Month 6: Sleep short of breath and headache | -44.44 (48.51)
  Month 6: Sleep Adequacy: number analyzed (Participants) | 39
  Month 6: Sleep Adequacy | 59.83 (81.33)
  Month 6: Sleep Somnolence: number analyzed (Participants) | 41
  Month 6: Sleep Somnolence | -18.15 (68.23)
  Month 6: Sleep Quantity (raw scores): number analyzed (Participants) | 37
  Month 6: Sleep Quantity (raw scores) | 30.17 (52.08)
  Month 6: Optimal Sleep Scale: number analyzed (Participants) | 7
  Month 6: Optimal Sleep Scale | -14.29 (37.80)
  Month 6: Sleep Problems Index I: number analyzed (Participants) | 41
  Month 6: Sleep Problems Index I | -29.01 (37.19)
  Month 6: Sleep Problems Index II: number analyzed (Participants) | 42
  Month 6: Sleep Problems Index II | -27.61 (37.60)
  Month 9: Sleep Disturbance: number analyzed (Participants) | 36
  Month 9: Sleep Disturbance | 4.54 (179.32)
  Month 9: Snoring: number analyzed (Participants) | 33
  Month 9: Snoring | -18.18 (52.02)
  Month 9: Sleep short of breath and headache: number analyzed (Participants) | 14
  Month 9: Sleep short of breath and headache | -57.14 (43.71)
  Month 9: Sleep Adequacy: number analyzed (Participants) | 34
  Month 9: Sleep Adequacy | 52.55 (113.18)
  Month 9: Sleep Somnolence: number analyzed (Participants) | 36
  Month 9: Sleep Somnolence | 7.55 (115.13)
  Month 9: Sleep Quantity (raw scores): number analyzed (Participants) | 33
  Month 9: Sleep Quantity (raw scores) | 9.33 (24.88)
  Month 9: Optimal Sleep Scale: number analyzed (Participants) | 9
  Month 9: Optimal Sleep Scale | -22.22 (44.10)
  Month 9: Sleep Problems Index I: number analyzed (Participants) | 36
  Month 9: Sleep Problems Index I | -13.61 (61.78)
  Month 9: Sleep Problems Index II: number analyzed (Participants) | 37
  Month 9: Sleep Problems Index II | -16.82 (49.82)
  Month 12: Sleep Disturbance: number analyzed (Participants) | 25
  Month 12: Sleep Disturbance | -16.56 (87.57)
  Month 12: Snoring: number analyzed (Participants) | 23
  Month 12: Snoring | -7.97 (81.28)
  Month 12: Sleep short of breath and headache: number analyzed (Participants) | 12
  Month 12: Sleep short of breath and headache | -58.33 (42.34)
  Month 12: Sleep Adequacy: number analyzed (Participants) | 21
  Month 12: Sleep Adequacy | 86.83 (142.51)
  Month 12: Sleep Somnolence: number analyzed (Participants) | 26
  Month 12: Sleep Somnolence | 0.59 (127.53)
  Month 12: Sleep Quantity (raw scores): number analyzed (Participants) | 24
  Month 12: Sleep Quantity (raw scores) | 22.50 (39.81)
  Month 12: Optimal Sleep Scale: number analyzed (Participants) | 5
  Month 12: Optimal Sleep Scale | -20.00 (44.72)
  Month 12: Sleep Problems Index I: number analyzed (Participants) | 26
  Month 12: Sleep Problems Index I | -19.99 (93.75)
  Month 12: Sleep Problems Index II: number analyzed (Participants) | 26
  Month 12: Sleep Problems Index II | -21.23 (66.11)

17. Secondary Outcome: Percentage Change From Baseline in Dermatology Life Quality-Index (DLQI) Score at Months 1, 3, 6, 9 and 12
Description: The DLQI was a 10-item participant-reported measure that rated how much a participant's skin problems had affected their life over the last week assigned to the following 6 dimensions: symptoms, daily life, leisure/sport, work/school, social life/relationship and treatment. Each question was scored from 0 to 3 where, 0=best quality of life and 3=greatest possible impairment of the quality of life (QoL). The total score was calculated as sum of scores and ranged from 0 (best QoL) to 30 (worst QoL), with higher scores indicating greater impairment of quality of life.
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Abrocitinib
Number analyzed (Participants) | 63
Percentage change
  Month 1 | -58.09 (33.22)
  Month 3: number analyzed (Participants) | 38
  Month 3 | -55.40 (54.83)
  Month 6: number analyzed (Participants) | 41
  Month 6 | -49.54 (73.27)
  Month 9: number analyzed (Participants) | 40
  Month 9 | -40.73 (85.53)
  Month 12: number analyzed (Participants) | 28
  Month 12 | -55.37 (70.83)

18. Secondary Outcome: Percentage Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Score at Months 1, 3, 6, 9 and 12
Description: HADS was a validated 14-item questionnaire to assess states of anxiety and depression. HADS consisted of 2 subscales: HADS-Anxiety (HADS-A) scale and HADS-Depression (HADS-D) scale, each of which comprised of 7 items among adults who were physically ill. Each item was rated on a 4-point scale, with scores ranging from 0 to 3, with 0 denoting lowest and 3 denoting highest anxiety or depression level. For both subscales the total score was derived by summing up the respective 7 items with total score ranging from 0 (no presence of anxiety and depression) to 21 (severe feeling of anxiety and depression); higher score indicated greater severity of anxiety and depression.
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Abrocitinib
Number analyzed (Participants) | 62
Percentage change
  Month 1: HADS anxiety score | -18.15 (43.84)
  Month 1: HADS depression score | -26.09 (55.72)
  Month 3: HADS anxiety score: number analyzed (Participants) | 37
  Month 3: HADS anxiety score | -25.67 (51.18)
  Month 3: HADS depression score: number analyzed (Participants) | 37
  Month 3: HADS depression score | -31.41 (78.54)
  Month 6: HADS anxiety score: number analyzed (Participants) | 40
  Month 6: HADS anxiety score | -19.24 (60.19)
  Month 6: HADS depression score: number analyzed (Participants) | 40
  Month 6: HADS depression score | -21.27 (75.52)
  Month 9: HADS anxiety score: number analyzed (Participants) | 37
  Month 9: HADS anxiety score | -17.88 (78.76)
  Month 9: HADS depression score: number analyzed (Participants) | 37
  Month 9: HADS depression score | -15.77 (89.51)
  Month 12: HADS anxiety score: number analyzed (Participants) | 26
  Month 12: HADS anxiety score | -32.25 (54.02)
  Month 12: HADS depression score: number analyzed (Participants) | 26
  Month 12: HADS depression score | -36.70 (58.61)

19. Secondary Outcome: Percentage Change From Baseline in EuroQol Five-dimensional-five Level (EQ-5D-5L) Score at Months 1, 3, 6, 9 and 12
Description: EQ-5D-5L was an instrument for measuring quality of life, including health benefits and health status on a visual analogue scale (VAS). EQ-5D health state profile has 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Responses to 5 dimensions comprise a health state/a single utility index value. E.g. if a participant responds "no problems" for each 5 dimensions, then health state was coded as "11111" with a predefined index value to it. Every health state (coded as combination of responses on each of 5 dimensions) has a unique predefined utility index value assigned to it, by EuroQol. Higher (positive) scores = better health state. The VAS component rates current health state on scale from 0 (worst imaginable health state) to 100 (best imaginable health state) ; higher scores indicate a better health state.
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Abrocitinib
Number analyzed (Participants) | 57
Percentage change
  Month 1: Index score | 26.76 (50.90)
  Month 1: VAS: number analyzed (Participants) | 56
  Month 1: VAS | 36.15 (51.76)
  Month 3: Index score: number analyzed (Participants) | 34
  Month 3: Index score | 29.86 (56.71)
  Month 3: VAS: number analyzed (Participants) | 36
  Month 3: VAS | 45.73 (54.75)
  Month 6: Index score: number analyzed (Participants) | 40
  Month 6: Index score | 30.36 (51.44)
  Month 6: VAS: number analyzed (Participants) | 38
  Month 6: VAS | 51.50 (60.27)
  Month 9: Index score: number analyzed (Participants) | 33
  Month 9: Index score | 25.37 (56.25)
  Month 9: VAS: number analyzed (Participants) | 34
  Month 9: VAS | 36.76 (43.67)
  Month 12: Index score: number analyzed (Participants) | 23
  Month 12: Index score | 32.44 (66.76)
  Month 12: VAS: number analyzed (Participants) | 23
  Month 12: VAS | 61.61 (63.38)

20. Secondary Outcome: Treatment Satisfaction Measured by Patient Benefit Index (PBI) at Months 1, 3, 6, 9 and 12
Description: PBI consisted of two one-sided questionnaires which were completed by participants before and after receiving a treatment. Total of 23 possible treatment goals were evaluated on importance scale from 0 ("not at all") to 4 ("very"). "Does not apply to me" was coded as "0". PBI was calculated by multiplying achieved benefits (respective PBI after baseline) with importance of the respective needs prior to therapy (PBI at baseline), dividing these products by sum of all importance items (PBI at baseline) and summing them up for all items. Total PBI score ranged from 0 (no benefit) to 4 (maximal benefit), where higher scores indicated more benefits. PBI questionnaire measured satisfaction at all points in time after baseline.
Time Frame: At Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abrocitinib
Number analyzed (Participants) | 64
Units on a scale
  Month 1 | 2.79 (0.99)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 2.92 (0.88)
  Month 6: number analyzed (Participants) | 42
  Month 6 | 3.12 (0.66)
  Month 9: number analyzed (Participants) | 37
  Month 9 | 2.92 (0.94)
  Month 12: number analyzed (Participants) | 29
  Month 12 | 3.07 (0.82)

21. Secondary Outcome: Number of Participants With Treatment Expectation Measured by PBI at Baseline
Description: PBI consisted of two one-sided questionnaires which were completed by participants before and after receiving treatment. Total of 25 possible treatment goals were evaluated on importance scale from 0 (" not at all") to 4 ("very"), where higher scores indicated more important goals. The responses to each treatment goal included: somewhat, moderately, quite, very, does not apply to me, not answered and not at all. Treatment expectation was measured at baseline.
Time Frame: At Baseline (Day 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Abrocitinib
Number analyzed (Participants) | 68
Participants
  Be free of pain: Somewhat | 2 [lower limit 0.82]
  Be free of pain: Moderately | 4 [lower limit 0.82]
  Be free of pain: Quite | 12 [lower limit 0.82]
  Be free of pain: Very | 45 [lower limit 0.82]
  Be free of pain: Does not apply to me | 5 [lower limit 0.82]
  Be free of pain: Not answered | 0 [lower limit 0.82]
  Be free of pain: Not at all | 0 [lower limit 0.82]
  Be free of itching: Somewhat | 0
  Be free of itching: Moderately | 2
  Be free of itching: Quite | 3
  Be free of itching: Very | 60
  Be free of itching: Does not apply to me | 0
  Be free of itching: Not answered | 3
  Be free of itching: Not at all | 0
  No longer have burning sensations on your skin: Somewhat | 0
  No longer have burning sensations on your skin: Moderately | 1
  No longer have burning sensations on your skin: Quite | 10
  No longer have burning sensations on your skin: Very | 54
  No longer have burning sensations on your skin: Does not apply to me | 2
  No longer have burning sensations on your skin: Not answered | 1
  No longer have burning sensations on your skin: Not at all | 0
  Be healed of all skin defects: Somewhat | 3
  Be healed of all skin defects: Moderately | 3
  Be healed of all skin defects: Quite | 12
  Be healed of all skin defects: Very | 49
  Be healed of all skin defects: Does not apply to me | 0
  Be healed of all skin defects: Not answered | 0
  Be healed of all skin defects: Not at all | 1
  Be able to sleep better: Somewhat | 5
  Be able to sleep better: Moderately | 5
  Be able to sleep better: Quite | 13
  Be able to sleep better: Very | 38
  Be able to sleep better: Does not apply to me | 6
  Be able to sleep better: Not answered | 0
  Be able to sleep better: Not at all | 1
  Feel less depressed: Somewhat | 4
  Feel less depressed: Moderately | 8
  Feel less depressed: Quite | 17
  Feel less depressed: Very | 31
  Feel less depressed: Does not apply to me | 8
  Feel less depressed: Not answered | 0
  Feel less depressed: Not at all | 0
  Experience a greater enjoyment of life: Somewhat | 2
  Experience a greater enjoyment of life: Moderately | 4
  Experience a greater enjoyment of life: Quite | 20
  Experience a greater enjoyment of life: Very | 37
  Experience a greater enjoyment of life: Does not apply to me | 5
  Experience a greater enjoyment of life: Not answered | 0
  Experience a greater enjoyment of life: Not at all | 0
  Have no fear that the disease will become worse: Somewhat | 4
  Have no fear that the disease will become worse: Moderately | 5
  Have no fear that the disease will become worse: Quite | 19
  Have no fear that the disease will become worse: Very | 36
  Have no fear that the disease will become worse: Does not apply to me | 3
  Have no fear that the disease will become worse: Not answered | 0
  Have no fear that the disease will become worse: Not at all | 1
  Be able to lead a normal everyday life: Somewhat | 2
  Be able to lead a normal everyday life: Moderately | 2
  Be able to lead a normal everyday life: Quite | 17
  Be able to lead a normal everyday life: Very | 44
  Be able to lead a normal everyday life: Does not apply to me | 3
  Be able to lead a normal everyday life: Not answered | 0
  Be able to lead a normal everyday life: Not at all | 0
  Be more productive in everyday life: Somewhat | 4
  Be more productive in everyday life: Moderately | 8
  Be more productive in everyday life: Quite | 11
  Be more productive in everyday life: Very | 39
  Be more productive in everyday life: Does not apply to me | 5
  Be more productive in everyday life: Not answered | 0
  Be more productive in everyday life: Not at all | 1
  Be less of a burden to relatives and friends: Somewhat | 5
  Be less of a burden to relatives and friends: Moderately | 11
  Be less of a burden to relatives and friends: Quite | 19
  Be less of a burden to relatives and friends: Very | 24
  Be less of a burden to relatives and friends: Does not apply to me | 9
  Be less of a burden to relatives and friends: Not answered | 0
  Be less of a burden to relatives and friends: Not at all | 0
  Be able to engage in normal leisure activities: Somewhat | 5
  Be able to engage in normal leisure activities: Moderately | 2
  Be able to engage in normal leisure activities: Quite | 14
  Be able to engage in normal leisure activities: Very | 41
  Be able to engage in normal leisure activities: Does not apply to me | 5
  Be able to engage in normal leisure activities: Not answered | 1
  Be able to engage in normal leisure activities: Not at all | 0
  Be able to lead a normal working life: Somewhat | 3
  Be able to lead a normal working life: Moderately | 5
  Be able to lead a normal working life: Quite | 15
  Be able to lead a normal working life: Very | 31
  Be able to lead a normal working life: Does not apply to me | 13
  Be able to lead a normal working life: Not answered | 0
  Be able to lead a normal working life: Not at all | 1
  Be able to have more contact with other people: Somewhat | 5
  Be able to have more contact with other people: Moderately | 9
  Be able to have more contact with other people: Quite | 19
  Be able to have more contact with other people: Very | 16
  Be able to have more contact with other people: Does not apply to me | 15
  Be able to have more contact with other people: Not answered | 0
  Be able to have more contact with other people: Not at all | 4
  Be comfortable showing yourself more in public: Somewhat | 4
  Be comfortable showing yourself more in public: Moderately | 9
  Be comfortable showing yourself more in public: Quite | 21
  Be comfortable showing yourself more in public: Very | 28
  Be comfortable showing yourself more in public: Does not apply to me | 5
  Be comfortable showing yourself more in public: Not answered | 1
  Be comfortable showing yourself more in public: Not at all | 0
  Be less burdened in your partnership: Somewhat | 3
  Be less burdened in your partnership: Moderately | 6
  Be less burdened in your partnership: Quite | 11
  Be less burdened in your partnership: Very | 30
  Be less burdened in your partnership: Does not apply to me | 17
  Be less burdened in your partnership: Not answered | 0
  Be less burdened in your partnership: Not at all | 1
  Be able to have a normal sex life: Somewhat | 3
  Be able to have a normal sex life: Moderately | 8
  Be able to have a normal sex life: Quite | 12
  Be able to have a normal sex life: Very | 27
  Be able to have a normal sex life: Does not apply to me | 13
  Be able to have a normal sex life: Not answered | 0
  Be able to have a normal sex life: Not at all | 5
  Be less dependent on doctor and clinic visits: Somewhat | 2
  Be less dependent on doctor and clinic visits: Moderately | 9
  Be less dependent on doctor and clinic visits: Quite | 19
  Be less dependent on doctor and clinic visits: Very | 37
  Be less dependent on doctor and clinic visits: Does not apply to me | 1
  Be less dependent on doctor and clinic visits: Not answered | 0
  Be less dependent on doctor and clinic visits: Not at all | 0
  Need less time for daily treatment: Somewhat | 3
  Need less time for daily treatment: Moderately | 9
  Need less time for daily treatment: Quite | 20
  Need less time for daily treatment: Very | 33
  Need less time for daily treatment: Does not apply to me | 2
  Need less time for daily treatment: Not answered | 0
  Need less time for daily treatment: Not at all | 1
  Have fewer out-of-pocket treatment expenses: Somewhat | 7
  Have fewer out-of-pocket treatment expenses: Moderately | 10
  Have fewer out-of-pocket treatment expenses: Quite | 12
  Have fewer out-of-pocket treatment expenses: Very | 30
  Have fewer out-of-pocket treatment expenses: Does not apply to me | 6
  Have fewer out-of-pocket treatment expenses: Not answered | 0
  Have fewer out-of-pocket treatment expenses: Not at all | 3
  Have fewer side effects: Somewhat | 2
  Have fewer side effects: Moderately | 7
  Have fewer side effects: Quite | 17
  Have fewer side effects: Very | 31
  Have fewer side effects: Does not apply to me | 10
  Have fewer side effects: Not answered | 0
  Have fewer side effects: Not at all | 1
  Find a clear diagnosis and therapy: Somewhat | 3
  Find a clear diagnosis and therapy: Moderately | 3
  Find a clear diagnosis and therapy: Quite | 14
  Find a clear diagnosis and therapy: Very | 42
  Find a clear diagnosis and therapy: Does not apply to me | 6
  Find a clear diagnosis and therapy: Not answered | 0
  Find a clear diagnosis and therapy: Not at all | 0
  Have confidence in the therapy: Somewhat | 2
  Have confidence in the therapy: Moderately | 2
  Have confidence in the therapy: Quite | 19
  Have confidence in the therapy: Very | 44
  Have confidence in the therapy: Does not apply to me | 1
  Have confidence in the therapy: Not answered | 0
  Have confidence in the therapy: Not at all | 0
  Get better skin quickly: Somewhat | 0
  Get better skin quickly: Moderately | 5
  Get better skin quickly: Quite | 9
  Get better skin quickly: Very | 54
  Get better skin quickly: Does not apply to me | 0
  Get better skin quickly: Not answered | 0
  Get better skin quickly: Not at all | 0
  Regain control of the disease: Somewhat | 2
  Regain control of the disease: Moderately | 3
  Regain control of the disease: Quite | 17
  Regain control of the disease: Very | 44
  Regain control of the disease: Does not apply to me | 1
  Regain control of the disease: Not answered | 0
  Regain control of the disease: Not at all | 1

22. Secondary Outcome: Number of Days With Topical Treatment Use
Description: Topical treatments included topical corticosteroids and topical calcineurin inhibitors. Number of days with topical treatment use was reported in this outcome measure. Number of days was calculated as date of first topical treatment - date of last topical treatment + 1.
Time Frame: Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Abrocitinib
Number analyzed (Participants) | 95
Days
  At Month 1 | 6.66 (10.12)
  At Month 3: number analyzed (Participants) | 83
  At Month 3 | 19.59 (31.57)
  At Month 6: number analyzed (Participants) | 66
  At Month 6 | 31.52 (52.98)
  At Month 9: number analyzed (Participants) | 52
  At Month 9 | 41.08 (71.48)
  At Month 12: number analyzed (Participants) | 42
  At Month 12 | 62.71 (97.25)

23. Secondary Outcome: Number of Days of Emollients Use
Description: Number of days with emollients use was calculated as: date of first emollients use - date of last emollients use + 1. The number of days with emollients use was reported in this outcome measure.
Time Frame: Months 1, 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Abrocitinib
Number analyzed (Participants) | 95
Days
  At Month 1 | 17.22 (14.41)
  At Month 3: number analyzed (Participants) | 83
  At Month 3 | 52.76 (43.39)
  At Month 6: number analyzed (Participants) | 66
  At Month 6 | 95.61 (74.54)
  At Month 9: number analyzed (Participants) | 52
  At Month 9 | 155.35 (105.94)
  At Month 12: number analyzed (Participants) | 42
  At Month 12 | 219.93 (135.11)

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) up to end of study (up to Month 12)
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. Event may be categorized as serious in 1 participant and non-serious in other, or participant may have experienced both serious and non-serious event. The safety analysis set consisted of all participants with informed consent who received at least one dose of abrocitinib.
Arm/Group | Abrocitinib
All-Cause Mortality (participants affected / at risk) | 0/112
Serious Adverse Events (participants affected / at risk) | 4/112
Other Adverse Events (participants affected / at risk) | 33/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abrocitinib (N=112)
Eczema herpeticum (Infections and infestations) | 1
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abrocitinib (N=112)
Nausea (Gastrointestinal disorders) | 14
Nasopharyngitis (Infections and infestations) | 11
Hyperlipidaemia (Metabolism and nutrition disorders) | 10
Headache (Nervous system disorders) | 6
Acne (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT05250115/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT05250115/SAP_001.pdf